CLINICAL TRIAL: NCT05613686
Title: Comparative Efficacy of Different Doses of Theta Burst Stimulation for Motor Recovery in Stroke Patients
Brief Title: Theta Burst Stimulation for Motor Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202204105DINB
Record Dates: First submitted 2022-10-30; First posted 2022-11-14 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Transcranial Magnetic Stimulation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- contralateral 1Hz+ipsilateral iTBS 1 (Experimental): Patients received contralateral 1 Hz and ipsilateral iTBS with protocol 1
  Interventions: Device: repetitive transcranial magnetic stimulation
- contralateral 1Hz+ipsilateral iTBS 2 (Experimental): Patients received contralateral 1 Hz and ipsilateral iTBS with protocol 2
  Interventions: Device: repetitive transcranial magnetic stimulation
- contralateral 1Hz (Active Comparator): Patients received contralateral 1 Hz and ipsilateral sham iTBS
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation technology. High and low frequencies of rTMS could modulate the excitability of the cerebral cortex. Theta burst stimulation (TBS) has achieved a similar effect to traditional rTMS mode. Intermittent TBS (iTBS) could upregulate cortical excitability of the primary motor cortex (M1) and continuous TBS (cTBS) with inhibitory effect.

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation technology. This study will compare efficacy of different doses iTBS in combination with inhibitory rTMS on motor recovery and cortical excitability in subacute stroke patients.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation technology.

High and low frequencies of rTMS could modulate the excitability of the cerebral cortex. Theta burst stimulation (TBS) has achieved a similar effect to traditional rTMS mode. Intermittent TBS (iTBS) could upregulate cortical excitability of the primary motor cortex (M1) and continuous TBS (cTBS) with inhibitory effect. Through modulating the excitability of bilateral hemispheres, rTMS could facilitate motor recovery in stroke patients.

This study will compare efficacy of different doses iTBS in combination with inhibitory rTMS on motor recovery and cortical excitability in subacute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.Unilateral ischemic or hemorrhagic stroke
* 2.Stroke within 3 months
* 3.Medical Research Council Scale for Muscle Strength in upper limb ≤ 3
* 4.No previous stroke, seizure, dementia, Parkinson's disease or other degenerative neurological diseases.
* 5.Patient could sit over 15 minutes
* 6.Age over 20

Exclusion Criteria:

* 1.Previous stroke, traumatic brain injury, brain tumor
* 2.With central nervous system disease (spinal cord injury, Parkinson's disease)
* 3.Any contraindication to rTMS (seizure, alcoholism, metal implant, pacemaker)
* 4.Patients unable to cooperate the treatment
* 5.Pregnancy
* 6.Depression

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-29 (Actual); Primary Completion 2024-10-29 (Estimated); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | 12 weeks post intervention
  Fugl-Meyer Assessment motor function set, score: 0-66, higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Medical Research Council (MRC) Scale for Muscle Strength | 1 week, 4 weeks, 12 weeks and 24 weeks post intervention
  Medical Research Council (MRC) Scale for Muscle Strength, assessing muscle strength from Grade 5 (normal) to Grade 0 (no visible contraction).
National Institutes of Health Stroke Scale | 1 week, 4 weeks, 12 weeks and 24 weeks post intervention
  National Institutes of Health Stroke Scale, The maximum possible score is 42, with the minimum score being a 0. Higher scores indicate a worse outcome.
Barthel Index | 1 week, 4 weeks, 12 weeks and 24 weeks post intervention
  Barthel Index, score 100-0. Higher scores indicate a better outcome.
Modified Rankin Scale | 1 week, 4 weeks, 12 weeks and 24 weeks post intervention
  Modified Rankin Scale, score from 0 to 6. Higher scores indicate a worse outcome.
MEP | 1 week, 4 weeks, 12 weeks and 24 weeks post intervention
  motor evoked potential
Fugl-Meyer Assessment | 1 week post intervention
  Fugl-Meyer Assessment motor function set, score: 0-66, higher scores indicate a better outcome.
Fugl-Meyer Assessment | 4 weeks post intervention
  Fugl-Meyer Assessment motor function set, score: 0-66, higher scores indicate a better outcome.
Fugl-Meyer Assessment | 24 weeks post intervention
  Fugl-Meyer Assessment motor function set, score: 0-66, higher scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ting Lin, M.D., Principal Investigator — The Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
will make further analysis

REFERENCES:
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449